CLINICAL TRIAL: NCT05464394
Title: Peroperative Administration of Tranexamic Acid in Roux-en-Y Gastric Bypass and One-anastomosis Gastric Bypass to Reduce Haemorrhage (PATRY Study): a Randomised Controlled Trial
Brief Title: Peroperative Administration of Tranexamic Acid in Roux-en-Y Gastric Bypass and One-anastomosis Gastric Bypass
Acronym: PATRY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Franciscus Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-031; 2022-001384-27 (EudraCT Number)
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Hemorrhage; Bleeding
Keywords: Gastric bypass; Tranexamic acid
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (Experimental): 1500mg Tranexamic acid
  Interventions: Drug: Tranexamic Acid Injection [Cyklokapron]
- Placebo (Placebo Comparator): sodium chloride
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Tranexamic Acid Injection [Cyklokapron] — A set dose of 1500 mg will be used, based on the study population with morbid obesity. It will be administered intravenous dissolved in 100 ml sodium chloride 0.9% in a time frame of 15-30 minutes, with a maximum of 100 mg/min.
  Arms: Tranexamic acid
Drug: Sodium chloride 0.9% — 100 ml sodium chloride 0.9% will be administered in a time frame of 15-30 minutes
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The incidence of bleeding after metabolic surgery seems to increase. The administration of a drug (tranexamic acid) that can reduce bleeding could possibly also reduce bleeding after metabolic surgery.

Objective: This study aims to determine whether administration of tranexamic acid before surgery can reduce postoperative bleeding in patients undergoing gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Primary metabolic procedure;
* Gastric bypass: Roux-en-Y gastric bypass or One-anastomoses gastric bypass;
* ≥18 years;
* Good command of the Dutch or English language.

Exclusion Criteria:

* Patients unwilling to give informed consent;
* Patients with a medical history of bleeding or VTE (defined as, pulmonary embolism (PE) or deep vein thrombosis (DVT));
* Patients who use anticoagulants;
* Arterial bleeding or (iatrogenic) bleeding during the procedure coming from surrounding organs or vascular structures such as the liver or the spleen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1524 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
re-intervention rate | 30 days
  To compare the re-intervention rate due to haemorrhage within 30 days postoperative, after peroperative administration of TXA versus placebo in patients receiving a RYGB or OAGB

SECONDARY OUTCOMES:
the use of haemostatic staple devices | peroperatively
  measurement (yes/no). Peroperatively, only on active bleeding a heamostatic staple device will be used. If there is no bleeding no haemostatic staple device will be used.
the use of fibrin sealant | peroperatively
  measurement (yes/no). Peroperatively, if the staple line is not actively bleeding but is oozing, fibrin sealant is used. If there is no oozing, fibrin sealant is not used.
blood loss | peroperatively
  blood loss in ml during surgery
haemoglobin decrease | 1 day
  haemoglobin decrease postoperative
heart rate increase | 1 day
  heart rate increase postoperative
number of suspicion on haemorrhage | 30 days
  number of suspicion on haemorrhage for which extra haemoglobin monitoring
number of suspicion on haemorrhage for which extra haemoglobin monitoring | 30 days
  number of suspicion on haemorrhage for which extra haemoglobin monitoring
VTE | 30 days
  VTE postoperative
complications rates | 30 days
  postoperative complications rates
length of hospital stay | 30 days
  length of hospital stay
duration of primary surgery | 1 day
  duration of primary surgery

IPD SHARING:
Plan to Share IPD: Yes
Data Statement: The identified individual clinical trial participant-level data, protocols, and the statistical analysis plan will be available upon reasonable request at publication. These data will be available for researchers who provide a methodologically sound proposal to achieve the aims in the approved proposal. Proposals should be directed to j.apers@franciscus.nl, and to obtain access, data requestors will need a data access agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Participant-level data, protocols, and the statistical analysis plan will be available upon reasonable request at publication. Within 1 year after the last follow-up.
Access Criteria: upon reasonable request

REFERENCES:
- [Derived] 't Hart JWH, Noordman BJ, Palsgraaf-Huisbrink J, Dunkelgrun M, Zengerink HF, Birnie E, van Det MJ, Boerma EG, de Castro SMM, Hazebroek EJ, Langenhoff BS, Verhoef C, Apers JA. Peroperative administration of tranexamic acid in Roux-en-Y and one-anastomosis gastric bypass to reduce haemorrhage in patients with morbid obesity: protocol for randomised controlled trial (PATRY trial). BMJ Open. 2024 May 6;14(5):e078853. doi: 10.1136/bmjopen-2023-078853. PMID 38719323